CLINICAL TRIAL: NCT01659567
Title: Prospective, Observational Study of Predictors of the Effectiveness of Pegylated Interferon in a Cohort of Patients With Hepatitis C in Georgia
Brief Title: A Study of Predictors of the Effectiveness of Pegylated Interferon in a Cohort of Participants With Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25544
Record Dates: First submitted 2012-07-27; First posted 2012-08-08 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Hepatitis C: Participants with chronic hepatitis C, treated with pegylated interferon alfa-2a (Pegasys) and ribavirin (Copegus) according to the current standard of care and in line with current summaries of product characteristics/local labelling, will be observed for up to 96 weeks.
  Interventions: Drug: Pegylated Interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon Alfa-2a — Pegylated interferon alfa-2a will be administered according to the current standard of care and in line with current summaries of product characteristics/local labelling.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin will be administered according to the current standard of care and in line with current summaries of product characteristics/local labelling.
  Other Names: Copegus

SUMMARY:
This prospective observational study will investigate predictive values of virological response in pegylated interferon alfa-2a (Pegasys)/ribavirin (Copegus) treatment-naive participants with chronic hepatitis C. Participants will be treated with pegylated interferon alfa-2a and ribavirin as prescribed by the physician. Data will be collected for a maximum of 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of chronic hepatitis C infection

Exclusion Criteria:

* Co-infection with human immunodeficiency virus (HIV) and/or hepatitis B
* Participants previously treated with pegylated interferon alfa-2a/ribavirin
* Participation in another clinical study within 30 days prior to study start of ML25544

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with chronic hepatitis C infection and naive to peginterferon/ribavirin treatment
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2011-04-06 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Georgia (3):
  - Hepatology Clinic Hepa, Tbilisi
  - Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - Ltd Mrcheveli, Tbilisi

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated Interferon Alfa-2a and Ribavirin: Participants with chronic hepatitis C, treated with pegylated interferon alfa-2a (Pegasys) and ribavirin (copegus) according to the current standard of care and in line with current summaries of product characteristics/local labelling, were observed for up to 96 weeks.
Period: Overall Study
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Started | 516
Completed | 393
Not Completed | 123
Not completed — Lack of Efficacy | 22
Not completed — Switched to Pegferon | 6
Not completed — Adverse Event | 12
Not completed — Good result at early stage of treatment | 5
Not completed — Withdrawal by Subject | 64
Not completed — Progression of the main disease | 1
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Population: Analysis population included all treated participants.
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.12 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 454

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response (SVR)
Description: SVR was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) level undetectable (less than [<] 15 international units per milliliter [IU/mL]) 24 weeks after completion of the actual treatment period (measured using the COBAS AmpliPrep [CAP]/ COBAS TaqMan [CTM] test). Percentage of participants achieving SVR was reported.
Time Frame: At 24 weeks after end of treatment (EOT) (up to 96 weeks), where EOT = up to 72 weeks
Population: Analysis population included all treated participants. Here, 'Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 225
percentage of participants | 79.1

2. Primary Outcome: Positive Predictive Value (PPV) of Rapid Viral Response (RVR) on SVR
Description: RVR was defined as HCV RNA less than or equal to (<=) 25 IU/mL at Week 4 using CAP/CTM test. The percentage of participants with probability that the participant who develops RVR would achieve SVR was termed as PPV of RVR on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: At 24 weeks after EOT (up to 96 weeks), where EOT = up to 72 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 185
percentage of participants | 93.1 [89.3 to 96.7]

3. Primary Outcome: PPV of Complete Early Viral Response (cEVR) on SVR
Description: cEVR was defined as HCV RNA <=25 IU/mL at Week 12, but not at Week 4 using CAP/CTM test. The percentage of participants with probability that the participant who develops cEVR would achieve SVR was termed as PPV of cEVR on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: At 24 weeks after EOT (up to 96 weeks), where EOT = up to 72 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
percentage of participants | 60.3 [48.3 to 72.3]

4. Secondary Outcome: Odds Ratio (OR) for Impact of Age on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of age (greater than [>] 42 years versus <=42 years) on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 225
odds ratio | 0.21 [0.10 to 0.47]

5. Secondary Outcome: OR for Impact of Gender on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of gender (male versus female) on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 225
odds ratio | 0.48 [0.13 to 1.69]

6. Secondary Outcome: OR for Impact of Body Weight on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of body weight on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 1.01 [0.99 to 1.02]

7. Secondary Outcome: OR for Impact of Baseline Level of Fibrosis (kPa) on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of baseline level of fibrosis on SVR. Level of fibrosis was measured in terms of kilopascals (kPa) using elastography. kPa score was categorized in 4 groups: 0 to 6.0; 6.1 to 9.9; 10.0 to 14.5; and 14.6 and above. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 186
odds ratio | 0.53 [0.38 to 0.74]

8. Secondary Outcome: OR for Impact of Baseline Alanine Transaminase (ALT) Level on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of baseline ALT level (>40 international units per liter [IU/L] versus <=40 IU/L) on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 215
odds ratio | 0.12 [0.02 to 0.92]

9. Secondary Outcome: OR for Impact of Baseline Viral Load Count on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of baseline viral load count (>800000 IU/mL versus <=800000 IU/mL) on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 219
odds ratio | 1.07 [0.56 to 2.03]

10. Secondary Outcome: OR for Impact of Overall Duration of Treatment on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of overall duration of treatment on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, EOT, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 1.05 [0.59 to 1.86]

11. Secondary Outcome: OR for Impact of Duration of Treatment After Achieving RVR on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of duration of treatment after achieving RVR (>18 weeks versus <=18 weeks) on SVR. RVR was defined as HCV RNA <=25 IU/mL at Week 4 using CAP/CTM test. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, Week 4, EOT, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 1.04 [0.92 to 1.18]

12. Secondary Outcome: OR for Impact of Duration of Treatment After Achieving cEVR on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of duration of treatment after achieving cEVR (>11 weeks versus <=11 weeks) on SVR. cEVR was defined as HCV RNA <=25 IU/mL at Week 12, but not at Week 4 using CAP/CTM test. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: Baseline up to 96 weeks (assessed at Baseline, Weeks 4, 12, EOT, 24 weeks after EOT [up to 96 weeks], where EOT = up to 72 weeks)
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 2.77 [1.14 to 6.72]

13. Secondary Outcome: OR for Impact of Cumulative Doses of Pegylated Interferon Alfa-2a on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of cumulative doses of pegylated interferon alfa-2a on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: At 24 weeks after EOT (up to 96 weeks), where EOT = up to 72 weeks
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 0.99 [0.99 to 1.00]

14. Secondary Outcome: OR for Impact of Cumulative Doses of Ribavirin on SVR
Description: The viral response development was assessed using univariate analysis with logistic regression model to calculate OR for impact of cumulative doses of ribavirin on SVR. SVR was defined as HCV RNA level undetectable (<15 IU/mL) 24 weeks after completion of the actual treatment period (measured using CAP/ CTM test).
Time Frame: At 24 weeks after EOT (up to 96 weeks), where EOT = up to 72 weeks
Population: Analysis population included all treated participants.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 516
odds ratio | 0.99 [0.99 to 1.00]

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks
Arm/Group | Pegylated Interferon Alfa-2a and Ribavirin
Serious Adverse Events (participants affected / at risk) | 17/516
Other Adverse Events (participants affected / at risk) | 256/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa-2a and Ribavirin (N=516)
Anemia (Blood and lymphatic system disorders) | 1
Anemia fourth degree (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia fourth degree (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia fourth degree (Blood and lymphatic system disorders) | 6
Hypoalbuminemia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Lingual bleeding (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Agitation (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Interferon Alfa-2a and Ribavirin (N=516)
Anemia (Blood and lymphatic system disorders) | 10
Bilirubinemia (Blood and lymphatic system disorders) | 2
Thyrotoxicosis second degree (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Thrombocytopenia second degree (Blood and lymphatic system disorders) | 1
Thrombocytopenia third degree (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 5
Leukopenia second degree (Blood and lymphatic system disorders) | 4
Leukopenia third degree (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 14
Neutropenia second degree (Blood and lymphatic system disorders) | 3
Neutropenia third degree (Blood and lymphatic system disorders) | 23
Liver enzymes incresed (ALT, AST other) (Blood and lymphatic system disorders) | 6
ST elevation (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Paresthesia (numbness in hands) (Cardiac disorders) | 1
Hemorrhoid varicose veins (Cardiac disorders) | 1
Hyperemia (Cardiac disorders) | 1
Flushing (Cardiac disorders) | 1
Alopecia/hair loss (Skin and subcutaneous tissue disorders) | 5
Itching/pruritus (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 6
Anal itching (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Herpes rash (Skin and subcutaneous tissue disorders) | 1
Left nostril furuncle (Skin and subcutaneous tissue disorders) | 1
Sweating - general (Skin and subcutaneous tissue disorders) | 1
Dry mouth (Skin and subcutaneous tissue disorders) | 3
Toxidermia (Skin and subcutaneous tissue disorders) | 1
Sty (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 65
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness in legs (Musculoskeletal and connective tissue disorders) | 1
Allergic reactions (Immune system disorders) | 8
Autoimmune thyroiditis (Immune system disorders) | 2
Headache (Nervous system disorders) | 31
Irritability (Nervous system disorders) | 8
Migraine (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Sexual potency impairment (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Flue-like syndrome (Respiratory, thoracic and mediastinal disorders) | 15
Sour throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 1
Abdominal pain upper/epigastric pain (Gastrointestinal disorders) | 3
Meteorism (flatulence) (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 128
Adynamy (General disorders) | 10
General weakness (General disorders) | 75
Rigors (General disorders) | 2
Sweating - general (General disorders) | 1
Blurred vision (Eye disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Earache (Ear and labyrinth disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Scalding during urination/urine scald (Renal and urinary disorders) | 1
Sexual potency impairment (Renal and urinary disorders) | 1
Weight decrease (Metabolism and nutrition disorders) | 1
Hyperthyroidism (Metabolism and nutrition disorders) | 4
Hypothyroidism (Metabolism and nutrition disorders) | 2
Loss of appetite (Metabolism and nutrition disorders) | 8
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 11
Emotional liability (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.